CLINICAL TRIAL: NCT02782689
Title: Evaluation of Efficacy and Safety of the 2-layer Compression System Kit Biflex® Versus the 4-layer Compression System PROFORE® in the Management of Venous Leg Ulcers (Stage C6).
Brief Title: Clinical Study to Assess Efficacy and Safety of a New Compression System in the Management of Venous Leg Ulcers
Acronym: COMPULCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in enrolling patients
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00287-40
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kit Biflex (Experimental): The Kit Biflex® will be applied according to manufacturer recommendations for 16 weeks or until full healing.
  Interventions: Device: Kit Biflex
- Profore (Active Comparator): The compression system Profore will be applied according to manufacturer recommendations for 16 weeks or until full healing.
  Interventions: Device: Profore

INTERVENTIONS:
Device: Kit Biflex — Two-layer reusable compression system
  Arms: Kit Biflex
Device: Profore — Four-layer compression system
  Arms: Profore

SUMMARY:
The primary objective of this study is to demonstrate the non-inferiority of the 2-layer compression system Kit Biflex® with regard of the 4-layer compression system PROFORE® in the treatment of venous leg ulcers in terms of complete healing at 16 weeks.

DETAILED DESCRIPTION:
This trial is a multicentre, randomized, comparative, open label clinical study conducted in vascular medicine centres in France, with 2 parallel groups of 100 patients each. The study will be conducted in patients suffering from venous leg ulcer (stage C6 of the CEAP classification for chronic venous disorders).

The patients will be randomised at the inclusion: they will receive with either Kit Biflex® or the reference device (Profore®) for maximum 16 weeks (or until full healing).

Investigator assessments are planned every 4 weeks +/- 3 days, for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients.
* Agreeing to wear a multilayer compression system throughout the study period.
* Presenting with an active venous leg ulcer: Duration between 1-24 months (whether a new ulcer or a recurrent ulcer); Surface area between 2-50 cm2; Venous, superficial or post-thrombotic ulcer confirmed by Doppler ultrasonography (dated within six months).
* With ankle circumference between 18-25 cm to allow the laying of the compression system.
* Able to follow the study instructions.
* Having read the information sheet and dated and signed the informed consent form.
* Covered by a health insurance system.

Exclusion Criteria:

* Scheduled surgery for the ulcer during the 16 weeks following inclusion.
* Clinical superinfected ulcer not controlled oral antibiotics.
* Malignant ulcer.
* Ulcer surface totally covered with dry fibrinous tissue or covered with black necrotic plaque on over 10% of its surface.
* Deep Vein Thrombosis within the last 3 months.
* Corticosteroids treatment (equivalent to more than 10 mg per day of prednisolone) ongoing or planned during the study.
* Radiotherapy, chemotherapy or immunosuppressive therapy ongoing or planned during the study.
* Erysipelas and lymphangitis.
* Lower extremity arterial disease or microangiopathy (Ankle Brachial Pressure Index <0.8 or> 1.3).
* Uncontrolled non-insulin dependent diabetes (HbA1c> 8%).
* Insulin-dependent diabetes.
* Confined to bed.
* With any uncontrolled severe and progressive disease.
* With a known or suspected hypersensitivity to any of the components of the study devices.
* Who had participated in a previous clinical study within the past 3 months.
* Pregnant women.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete wound closure (100% re-epithelialisation) over the treatment period | 16 weeks
Nature and frequency of adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc GILLET, MD, Principal Investigator
Locations (1):
- Thuasne, Levallois-Perret, France